CLINICAL TRIAL: NCT01015456
Title: The Clinical Efficacy and Economic Evaluation of EC-MPS (Myfortic) in the Treatment of Relapse or Resistant Proliferative Lupus Nephritis
Brief Title: The Efficacy of Enteric-coated Mycophenolate Sodium (EC-MPS) (Myfortic) in The Treatment of Relapse or Resistant Proliferative Lupus Nephritis
Acronym: CONTROL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data Safety Monitoring Board concerning of the participants' safety
Sponsor: Chulalongkorn University (Other)
Collaborators: Clinical Research Collaborative Network (Network); Health Intervention and Technology Assessment Program (HITAP) (Unknown)
Responsible Party: Principal Investigator, Yingyos Avihingsanon, Associate Professor., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-001; Lupus Research Unit; CRCN; HITAP
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; mycophenolate sodium; cyclophosphamide
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral mycophenolate sodium 1440 mg per day for 12 months
  Interventions: Drug: mycophenolate sodium
- 2 (Active Comparator): Intravenous cyclophosphamide monthly for 6 months
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: mycophenolate sodium — per oral, twice daily, for 12 months
  Other Names: Myfortic
  Arms: 1
Drug: cyclophosphamide — intravenous, monthly, for 6 months
  Other Names: Cytoxan
  Arms: 2

SUMMARY:
To investigate the efficacy and safety of enteric-coated mycophenolate sodium (Myfortic) as compared to intravenous cyclophosphamide in the treatment of active nephritis. The primary outcomes are complete and partial renal remission, as assessed by renal function, urinary sediment and proteinuria in patients with International Society of Nephrology/ Renal Pathology Society (ISN/RPS) class III or IV lupus nephritis.

DETAILED DESCRIPTION:
In this study, there are two sub-studies in order to define secondary endpoints.

1. Pharmacokinetics study of Mycophenolic acid
2. Identify biomarkers for therapy-resistant prediction.
3. Identify biomarkers for predicting a loss of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* age 16 years of above at the time of screening
* ability and willingness to provide written informed consent (or to obtain consent from parent guardian where applicable) and to comply with the schedule of protocol requirements
* Diagnosis of SLE according to ACR criteria. At least 4 criteria must have been present for the diagnosis of SLE. The 4 criteria do not have to be present at the time of screening
* Active lupus nephritis defined as follows: Biopsy proven (within 16 weeks prior to screening) ISN Class III or IV (A or A/C) not include III(C) IV(C) and VI (>90% chronic irreversible scarring)
* Relapse or resistant to (3 consecutive doses) IVCY
* Resistant lupus or Relapse lupus nephritis defined as follows:

  * Increase in serum creatinine >/= 0.3 mg/dl or
  * Increase in proteinuria > 1.5 g/day (which must have improved by ≥ 50% in the preceding 3 months)
* Life-time cumulative dose of IVCY > 6 grams
* Female patients of childbearing potential must have a negative serum pregnancy

Exclusion Criteria:

Relates to SLE

* Diagnosis of rapid progressive glomerulonephritis (RPGN): doubling serum creatinine and/or crescentic glomeruli ≥ 30%
* Severe renal impairment as defined by calculated creatinine clearance or MDRD-GFR < 30 ml/min(except creatinine clearance or MDRD-GFR > 50 ml/min in the 12 weeks prior to screening)
* History of serious disease or complication in any organ system that not appropriate to treatment immunosuppressive drug groups.
* Severe extra-renal organ involvement

Related to Treatment

* Previous of any Mycophenolate groups in the 6 months prior to screening
* Treatment with any investigational drugs in the 3 months prior to screening

Related to General Health

* Pregnancy or breast feeding mothers.
* Concomitant condition which has required treatment moderate to high dose steroid in the 12 weeks prior to screening.
* Evidence of significant uncontrolled concomitant disease in any organ system not related to SLE.
* History of cancer, including solid tumors, hematological malignancies and carcinoma.
* Evidence of current abuse of drugs or alcohol.

Related to Laboratory Findings

* Neutrophile < 1,500/mm3, Hb < 7g/L, Platelet < 50,000/mm3 (except active SLE)
* Positive HBsAg or anti-HCV or anti-HIV.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of enteric-coated Mycophenolate Sodium at 12 months in the treatment of lupus nephritis | 12 months

SECONDARY OUTCOMES:
The cost-effectiveness of using enteric-coated Mycophenolate Sodium as compared to standard treatment | 12 months
The ratio of patients with declined renal function | 12 months
Time to remission | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yingyos Avihingsanon, MD, Principal Investigator — Chulalongkorn University
Locations (3):
- Thailand (3):
  - Khon Kaen University, Khon Kaen, Changwat Khon Kaen
  - Nopparat Rajathani, Bangkok
  - Thammasart University, Pathum Thani

REFERENCES:
- [Derived] Anutrakulchai S, Panaput T, Wongchinsri J, Chaishayanon S, Satirapoj B, Traitanon O, Pima W, Rukrung C, Thinkhamrop B, Avihingsanon Y. A multicentre, randomised controlled study of enteric-coated mycophenolate sodium for the treatment of relapsed or resistant proliferative lupus nephritis: an Asian experience. Lupus Sci Med. 2016 Jan 14;3(1):e000120. doi: 10.1136/lupus-2015-000120. eCollection 2016. PMID 26835147
- See also: Lupus Research Unit — http://www.lupus.research.chula.ac.th/